CLINICAL TRIAL: NCT03747198
Title: The Effects of Methylsulfonylmethane on Knee Laxity in Active Young Females
Brief Title: Methylsulfonylmethane on Knee Laxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Bergstrom Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1356922
Record Dates: First submitted 2018-11-09; First posted 2018-11-20 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Ligament Injury; Ligament; Laxity; Tendon Rupture; Tendon Injuries
MeSH Terms: conditions — Joint Instability; Tendon Injuries | interventions — dimethyl sulfone

STUDY DESIGN:
Intervention Model Description: double blinded randomized parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: MSM tablets will be packaged and labelled (intervention A or B) by Bergstrom nutrition off-site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methylsulfonylmethane (Experimental): Subjects will be given 2 g/day of methylsulfonylmethane (MSM). Salivary estrogen will be measured around ovulation and menstruation each month for 3 months. Knee laxity will be measures 2 times per month at the same time points (ovulation, menstruation).
  Interventions: Dietary Supplement: methylsulfonylmethane
- Placebo (Placebo Comparator): Subjects will be given 2 g/day placebo (rice flour). Salivary estrogen will be measured around ovulation and menstruation each month for 3 months. Knee laxity will be measures 2 times per month at the same time points as the intervention arm (ovulation, menstruation).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: methylsulfonylmethane — Subjects will be given 2 g/day methylsulfonylmethane.
  Other Names: MSM
  Arms: methylsulfonylmethane
Other: Placebo — Subjects will be given 2 g/day placebo (rice flour).
  Arms: Placebo

SUMMARY:
The proposed research will focus on determining the effect of methylsulfonylmethane (MSM) on knee laxity changes through the menstrual cycle in young active females.

As an extension to recent discovery, that MSM reverses the negative effect of estrogen on engineered ligament function, the proposed work is designed to determine whether MSM can decrease the negative effect of estrogen on knee laxity in females.

Ligament function is determined by the content and cross-linking of collagen, which is influenced by a milieu of biochemical and mechanical parameters. The greater the amount and cross-linking the greater the stiffness and strength of these connective tissues. In engineered ligaments it has been previously shown that the high levels of estrogen, normally present in the days before and after ovulation, can inhibit the cross-linking enzyme lysyl oxidase. This decrease in collagen cross-linking likely increases connective tissue laxity and contributes to observed 4-fold greater occurrence of anterior cruciate ligament (ACL) rupture in females. Conversely, MSM increases collagen cross-linking and recent work conducted by the Baar lab in engineered human ligaments treated with high estrogen demonstrated that MSM could completely reverse the effects of estrogen on ligament mechanics.

The proposed research aims to advance this promising pre-clinical data and apply in a clinical trial. This research also proposes to quantify that knee laxity increases up to 5mm between the first day of menstruation and the day after ovulation and also that the magnitude of the increase in laxity is directly related to the magnitude of the change in estrogen. Importantly, a direct relationship between knee laxity and ACL rupture exists. For every 1.3mm increase in anterior-posterior knee displacement, the odds of ACL rupture increase 4-fold. Therefore, any treatment that decreases knee laxity could be expected to reduce ACL ruptures and have widespread application across the general active population and high-level athletics.

DETAILED DESCRIPTION:
Familiarization: Subjects would come to the Human Performance lab for a study orientation to be informed of the goals of the study, have anthropometric data collected (InBody770, In Body, Cerritos, CA) and familiarized with all testing and data collection tools. The purpose of this is to collect anthropometric data, review the study procedures and study requirements.

Determination of menstruation date: After study familiarization instructions will be given to contact the research team and come back to the lab on the first day of menstruation to establish the individual study timeline. An ovulation kit will be provided. The ovulation kit would then be started at the end of the first reported menstrual cycle and be used daily until the 2-4 days of high estrogen (ovulation) are established.

Baseline data: After menstruation date is established, for the first two months of the study, subjects would come to the lab on the first day of menstruation and the day after ovulation, have their knee laxity measured (GNRB dynamic laximeter, Prothia, Worcester, MA) and salivary analysis to determine estrogen levels. The first two months would determine normal changes in knee laxity and estrogen levels throughout the cycle within each subject.

Intervention: Following the second ovulation testing day and once baseline values are established, subjects would be provided with 3 months of MSM or placebo control (rice flour) and instructed to take 2g each morning for the subsequent 3 months. Month 3 would serve as an MSM loading month and subjects would return to the laboratory throughout months 4 and 5 (day 14 and first day of menstruation) for mechanical and estrogen testing.

MSM or placebo treatments: The study will be a randomized double-blinded placebo-controlled trial. MSM or placebo capsules would be provided in a double blinded manner following the second mechanical test. Each individual would consume 2g of either the MSM or placebo control for the remainder of the study.

Intervention Product and Preparation Intervention: MSM (OptiMSM®) is a pure, generally recognized as safe (GRAS) designated product. MSM can be found in small amounts in corn, tomatoes, tea, coffee, milk.

Placebo: Rice flour is a commonly ingested food or additive. Intervention and placebo will be encapsulated in 1g vegetarian capsules (Hypromellose Capsule).

Both intervention and placebo capsules are identically transparent with white powder inside. Capsules containers with 805 capsules (2g per day for each month plus extra) will be prepared, packaged by Bergstrom nutrition and transported with blinded code (A or B) so only individuals responsible for intervention and placebo preparation are removed from conducting the study and are off site (Vancouver, Washington).

Product will be labelled by Bergstrom Nutrition. Subject ID and month (3, 4, or 5) will be filled in manually by University of California, Davis researcher upon randomization.

Determination of knee laxity: Knee laxity will be determined using a GNRB dynamic laximeter following established protocols. Briefly, with the femur held in place, a controlled pressure will be applied to the calf. The pressure increases from 0 to 200 Newtons and a sensor measures kneecap displacement (laxity) in millimeters.

Determination of estrogen levels: Salivary samples will be taken on the first day of menstruation and one day following ovulation for the 4 months of testing (month 1, 2, 4, 5). Estradiol levels in the saliva will be determined using the Estradiol Saliva ELISA kit (Rocky Mountain Diagnostics, CO) as per manufacturer's instructions.

Data Collected:

* Record of menstrual cycle
* Salivary estradiol levels as described above
* Measurements of knee laxity

ELIGIBILITY:
Inclusion Criteria:

* • Regular menstrual cycle (~1 x month)

  * Not using oral contraceptive
  * No history of serious knee injury (e.g. ACL rupture)
  * Not currently pregnant (known)
  * Not routinely taking medication or supplements that would interact with study measures or be contraindicated (e.g. steroid injections)

Exclusion Criteria:

* • Irregular menstrual cycling (1 x month)

  * Using oral contraceptive
  * History of serious knee injury (e.g. ACL rupture)
  * Currently pregnant or potential of being pregnant
  * Routinely taking medication or supplements that would interact with study measures or be contraindicated (e.g. steroid injections)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female menstruate and the study is base on hormonal fluctuations that happen concurrent to the menstrual cycle and the effects of estrogen on knee laxity. This is why the study is including only females.
Enrollment: 32 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Kneecap displacement (i.e. knee laxity) | 5 months
  Knee laxity will be measured at months 4 and 5 after the 3-month intervention period of the study. The measurement will be made in millimeters using a specially designed GNRB arthrometer, which is a computerized and automatic medical device developed and validated by Genourob.

SECONDARY OUTCOMES:
Weight | 1 day
  The subjects weight (kg) will be commented at the start of the study for subject demographic purposes. Measurements will be made with the InBody 570 Body Composition analyzer.
Height | 1 day
  The subjects height (cm) will be commented at the start of the study for subject demographic purposes. Measurements will be made with a stadiometer.
Body composition | 1 day
  The subjects body composition (% body fat) will be commented at the start of the study for subject demographic purposes. Measurements will be made with the InBody 570 Body Composition analyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurobiology, Physiology & Behaviour, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No